CLINICAL TRIAL: NCT00000426
Title: Treatment of Calcium Deficiency in Young Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AR042155 (NIH); R01AR042155 (NIH); NIAMS-005
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Osteoporosis
Keywords: Calcium deficiency; Dietary calcium; Dietary protein; Osteoporosis; Calcium supplement; Bone density; Bone mass; Bone mass accumulation
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: Calcium supplement

SUMMARY:
This study looks at the effects of calcium supplementation on bone density in women in their third decade of life. We placed women aged 19-27 who take in low amounts of calcium in their diets in one of two groups. We will give women in one group a placebo (inactive pill) and women in the other group 1500 milligrams of calcium per day (as calcium carbonate). We will monitor the results by looking at the change in bone mineral density measured at the hip, total body, forearm, and spine. Treatment will last 3 years.

DETAILED DESCRIPTION:
This is a randomized, controlled trial of calcium carbonate supplementation (1500 milligrams per day) in third-decade women with low calcium-to-protein intakes. We accept women aged 19-27 on the basis of good health and the 7-day food diary demonstrating a dietary calcium-to-protein ratio (in milligrams:grams) that does not exceed 13. The outcome variable is the change in BMD at hip, total body, forearm, and spine. Treatment lasts for 3 years. We expect that bone mass will increase in both groups but will increase to a greater extent in the calcium-supplemented group than in the nonsupplemented group.

ELIGIBILITY:
Inclusion Criteria:

* Women in good health
* Dietary calcium-to-protein ratio (in mg:g, as assessed by 7-day food diary) does not exceed 13

Exclusion Criteria:

* Smoking
* Pregnancy
* Lactation
* Endocrine disease

Ages: 19 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Start 1995-01; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Heaney, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Background] Heaney RP. Phosphorus nutrition and the treatment of osteoporosis. Mayo Clin Proc. 2004 Jan;79(1):91-7. doi: 10.4065/79.1.91. PMID 14708952